CLINICAL TRIAL: NCT06692283
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Denifanstat in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease (MALSD)/Metabolic Dysfunction-Associated Steatohepatitis (MASH)
Brief Title: A Phase 3 Study Evaluating the Safety and Efficacy of Denifanstat in Patients With MASLD and MASH
Acronym: FASCINIT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB2640-CLIN-011
Record Dates: First submitted 2024-09-10; First posted 2024-11-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: MASLD; MASH; NASH; Metabolic Dysfunction-Associated Steatotic Liver Disease; Metabolic Dysfunction-Associated Steatohepatitis; Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver
Keywords: fatty liver; steatohepatitis; steatotic liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — TVB-2640

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Denifanstat 50 mg (Experimental): Denifanstat tablet, orally, once daily
  Interventions: Drug: denifanstat
- Placebo (Placebo Comparator): Placebo tablet, orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: denifanstat — Tablet
  Other Names: TVB-2640
  Arms: Denifanstat 50 mg
Drug: Placebo — Matching tablet
  Arms: Placebo

SUMMARY:
A phase 3, randomized, double-blind, placebo-controlled study evaluating the safety and tolerability of denifanstat 50 mg compared to placebo in patients with metabolic dysfunction-associated steatotic liver disease (MALSD)/metabolic dysfunction-associated steatohepatitis (MASH) after 52 weeks of treatment.

DETAILED DESCRIPTION:
Up to 2000 patients will be randomized to receive either denifanstat 50 mg or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to participate in the study and provide written informed consent.

2. Adults between 18 and 75 years of age.

3. Body mass index (BMI) ≥23 kg/m2 for Asian patients and ≥25 kg/m2 for patients of other races.

4. Presence of metabolic risk factor(s), as follows:

1. T2DM

   OR
2. At least 2 out of 4 of the following:

   * BMI ≥30 kg/m2,
   * Hypertension, or on active antihypertensive treatment
   * Elevated fasting serum TGs or on active treatment for hypertriglyceridemia
   * Reduced fasting serum HDL-c, or on active treatment for dyslipidemia.

5. For patients with T2DM:

1. HbA1c ≤9.5%
2. If treatment naive: patients must have been diagnosed for at least 12 weeks prior to screening

6. Suspected or confirmed diagnosis of MASH or MASLD or non-invasively diagnosed MASH or MASLD

7. Stable ALT and AST levels

Exclusion Criteria:

1. Previous intake of an approved MASH medication

2. Exclusionary laboratory values:

1. ALT and/or AST >5 × ULN.
2. ALP ≥2 × ULN.
3. Total serum bilirubin concentration >1.3 mg/dL.
4. Serum albumin concentration <3.5 g/dL.
5. International normalized ratio (INR) >1.3, except for patients receiving anticoagulant treatment.
6. Platelet count <140,000/μL.
7. Fasting TG level ≥500 mg/dL.
8. eGFR <45 mL/min/1.73 m2.

3. History of excessive alcohol intake for a period of more than 3 consecutive months within 1 year prior to screening.

4. Presence of cirrhosis on liver histology and/or cross-sectional imaging evidence consistent with cirrhosis and/or portal hypertension.

5. Current or historical clinically evident hepatic decompensation.

6. Evidence of another form of active liver disease.

7. Positive serologic evidence of current infectious liver disease.

8. MELD score ≥12.

9. Planned or history of liver transplantation.

10. Prior or planned bariatric surgery.

11. Gain or loss of >5% of body weight in the 3 months or >10% of body weight in the 6 months prior to screening, qualifying liver biopsy, and the baseline visit (V1).

12. Any of the following conditions or procedures within 6 months prior to the baseline visit (V1):

1. Myocardial infarction
2. Cardiac revascularization surgery
3. Unstable angina
4. Transient ischemic attack, stroke, or cerebrovascular disease

13. Unstable or undiagnosed arrhythmias.

14. Uncontrolled high BP.

15. Malignancy with a complete remission date within 5 years prior to the baseline visit (V1).

16. Any current or history of hepatocellular carcinoma.

17. Diabetes other than T2DM

18. Uncontrolled hypothyroidism.

19. Any other known serious disease or other disease which in the Investigator's opinion would exclude the patient from participating in the study.

20. Use of a nonpermitted concomitant medication within 30 days or 5 half-lives prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome Measure: TEAEs | 52 weeks
  Incidence of treatment-emergent adverse events (TEAEs) in patients with MASLD/MASH treated with denifanstat 50 mg compared to placebo after 52 weeks of treatment.

IPD SHARING:
Plan to Share IPD: No